CLINICAL TRIAL: NCT06158789
Title: Single-center, Open, Prospective, Single-arm, Feasibility, Investigator-initiated Trial for Assessment of Efficacy and Safety of Repetitive Blood Brain Barrier Disruption Using High Intensity Focused Ultrasound 'ExAblate 4000 Type 2' in Patients With Alzheimer's Disease
Brief Title: Repetitive Blood Brain Barrier Opening for Alzheimer's Disease.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kyung Won Chang (Other)
Collaborators: Yonsei University (Other)
Responsible Party: Sponsor-Investigator, Kyung Won Chang, Clinical professor, Severance Hospital
Organization: Severance Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YUSHAD-02
Record Dates: First submitted 2023-11-20; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Focused ultrasound treatment group (Experimental)
  Interventions: Procedure: MR guided low intensity focused ultrasound

INTERVENTIONS:
Procedure: MR guided low intensity focused ultrasound — Low intensity focused ultrasound opens the blood brain barrier

SUMMARY:
This study was focused on comparing the efficacy of repetitive Focused ultrasound mediated BBB opening in alzhemer's disease in increased number of treatment session and shorter intervals.

ELIGIBILITY:
Inclusion Criteria:

* Age over 50 to 85
* MMSE below 23
* FBB-PET positive
* FDG-PET shows alzheimer -induced neurodegeneration
* Dementia or cognitive impairment due to alzhemer's disease
* participants who have taken over 3 months of medication related with cognitive improvement
* Someone who can express their sensations during the procedure.
* Individuals who have voluntarily decided to participate in this clinical trial and have provided written consent on the informed consent form.
* Individuals with a commitment to adhere to the clinical trial protocol.

Exclusion Criteria:

* If any of the following exclusion criteria apply, participation in this clinical trial is not allowed.

If the severity score for the items "Delusions," "Hallucinations," or "Agitation/Aggression" in the CGA-NPI (Caregiver-Administrated Neuropsychiatry Inventory) test is greater than 2.

Note: Since the CGA-NPI requires the patient's caregiver to complete the survey, the caregiver must be present during the questionnaire.

Individuals with sensitivity/allergy or contraindications to the MRI contrast agents Gadolinium (Gadovist®) or ultrasound contrast agent Definity.

Contraindications:

Gadolinium (Gadovist®): Patients with untreated hypokalemia. Definity: Patients who have undergone right-left shunt, bidirectional shunt, or temporary right-left shunt, patients scheduled to undergo extracorporeal shock wave lithotripsy within 24 hours, clinically unstable or worsening congestive heart failure patients, acute myocardial infarction or acute coronary syndrome patients, patients at high risk of arrhythmias due to severe ventricular arrhythmias or prolongation of the QT interval, patients showing signs and symptoms of carbon dioxide retention or hypoxemia, patients with conditions that may induce pulmonary artery hypertension due to severe pulmonary insufficiency, severe pulmonary fibrosis, or damage to the pulmonary artery structure.

Individuals with standard contraindications to MR imaging, including the presence of metal devices incompatible with MRI.

Individuals with sensitivity/allergy or contraindications to anesthetic agents used for conscious sedation during procedures where conscious sedation is required.

Individuals with any of the following findings in the MRI examination:

Severe ischemic changes (Fazeka criteria score > 2, Lacunes count > 5, or Cerebral microbleeds count > 3).

Active or chronic infection/inflammation. Acute or chronic bleeding. Tumor/space-occupying lesion. Meningeal enhancement. Intracranial hypotension.

Individuals with more than 30% of the skull area through which the sonication (Sonication) path passes covered with scars, scalp disorders (e.g., eczema), or atrophied scalp.

Individuals with a history of seizure disorder or epilepsy that could be exacerbated due to blood-brain barrier opening.

Individuals with a history of bleeding disorders.

Individuals with severe cardiac conditions or unstable hemodynamic status (e.g., uncontrollable hypertension, arrhythmias, angina, etc.).

Individuals with impaired kidney function (Glomerular filtration rate < 30 mL/min/1.73 m²).

Individuals with severe brain atrophy to an extent that cannot be targeted.

Individuals who are HIV (Human Immunodeficiency Virus) positive and have a high likelihood of developing HIV encephalitis as HIV enters the brain parenchyma.

Individuals with potential vascular-origin infections that can enter the brain parenchyma, leading to meningitis or brain abscess.

Individuals with a thin blood-brain barrier, known to have homozygosity of the Apolipoprotein E allele (ApoE4).

Pregnant or lactating women.

For fertile women*, those who have agreed to use clinically appropriate contraceptive methods** during the trial period.

Definition of fertile women: Women who have experienced menarche and are not defined as postmenopausal after 12 months of amenorrhea without any surgical infertility procedures (e.g., hysterectomy or bilateral oophorectomy).

** Clinically appropriate contraceptive methods: For women, it is defined as "[Intrauterine device (e.g., loop, Mirena), chemical contraception (birth control pills), or subcutaneous contraceptive devices (e.g., Implanon)] + Physical contraceptive methods (male or female)," and for tubal ligation or laparoscopic contraception (a type of tubal ligation).

Individuals currently participating in another clinical trial or who have participated in another clinical trial within 90 days of the screening date.

Other cases where the investigator deems participation in the clinical trial inappropriate due to ethical or potential impact on clinical trial results.

Specific reasons should be documented in the case record.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2024-01-19 (Estimated)

PRIMARY OUTCOMES:
Changes in Standard Uptake Value Ratios (SUVR) on FBB-PET | Screening, 2weeks after final procedure
  Conducting FBB (18F-Florbetaben)-PET scans to confirm the presence of Amyloid beta protein (Aβ) plaques in the brain, the study compares and analyzes the global and regional standard uptake value ratios (SUVR) before the first procedure (Visit 1) and after the third procedure (Visit 12). The cerebellar gray matter is used as a reference region, and the analysis includes whole-brain as well as regional (Frontal/Temporal) SUVR.
Changes in CGA-NPI (Caregiver-administered neuropsychiatric inventory) Scores and Percentage Change | Screening, 2weeks after every session, 2months after final session
  To assess the cognitive function of participants, the CGA-NPI (Caregiver-Administered Neuropsychiatric Inventory) test is administered before the first procedure (Visit 1) and compared to scores after the first, second, and third procedures (Visits 4, 8, 12, 13). Changes in CGA-NPI scores and percentage changes (%) are investigated at each assessment point, with responses provided by the same participant's caregiver. Higher scores indicate severity of neuropsychiatric symptoms and 0 indicates no symptom.
Changes in K-MMSE(Korean version of Mini Mental State Exam) Test Scores and Percentage Change | Screening, 2months after final session
  For evaluating cognitive function, the K-MMSE (Korean version of Mini Mental State Exam) test is conducted before the first procedure (Visit 1) and compared to scores after the third procedure (Visits 12, 13). Changes in K-MMSE scores and percentage changes (%) are examined. Higher scores indicate better cognition.
Changes in SNSB(Seoul Neuropsychological Screening Battery)Test Scores and Percentage Change | Screening, 2months after final session
  Assessing cognitive function, the SNSB (Seoul Neuropsychological Screening Battery) test is performed before the first procedure (Visit 1) and compared to scores after the third procedure (Visit 13). Changes in SNSB scores and percentage changes (%) are investigated. Higher scores indicate better cognition.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Woo Chang, MD,PhD, Principal Investigator — Yonsei University; Byoung Seok Ye, MD,PhD, Study Chair — Yonsei University; Kyung Won Chang, MD, Study Director — Yonsei University; Kyung Won Chang, MD,PhD, Study Director — Yonsei University
Locations (1):
- Yonsei University Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park SH, Baik K, Jeon S, Chang WS, Ye BS, Chang JW. Extensive frontal focused ultrasound mediated blood-brain barrier opening for the treatment of Alzheimer's disease: a proof-of-concept study. Transl Neurodegener. 2021 Nov 5;10(1):44. doi: 10.1186/s40035-021-00269-8. PMID 34740367